CLINICAL TRIAL: NCT04398979
Title: Minimally Invasive Surgical Ablation for Standalone Atrial Fibrillation
Brief Title: Surgical Ablation for Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Investigator of the First Hospital of Nanjing Medical University, Nanjing Medical University
Other Study IDs: JPSH-AF2012
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Thoracoscopic Atrial fibrillation Ablation — After blunt dissection of the oblique and transverse sinus, an AtriCure Lumitip Dissector was introduced around the pulmonary veins. Pulmonary vein isolation was achieved with an AtriCure Isolator Synergy ablation clamp around the pulmonary vein antrum at least six times for each side. Ganglionated plexus identification and ablation were performed using an AtriCure Synergy ablation pen. The additional superior and inferior ablation lines connecting the bilateral pulmonary vein isolations were created by applying the AtriCure Synergy ablation pen. Following completion of the ablation on the right side, ablation on the left side was accomplished in a similar manner. The ligament of Marshall was dissected by electrical cautery. Conduction block was confirmed upon completion of the ablation procedure on the left side.

SUMMARY:
Minimally invasive approaches for surgical treatment have been advocated as a treatment option for stand-alone atrial fibrillation (AF). This study will investigate the clinical outcomes after minimally invasive surgical ablation of both paroxysmal and persistent/longstanding persistent AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) patients with a previous stroke are often at a high risk of recurrent stroke and bleeding. Minimally invasive approaches for surgical treatment have been advocated as a treatment option for stand-alone AF. This study will investigate the clinical outcomes after minimally invasive surgical ablation of both paroxysmal and persistent/longstanding persistent AF. Neurological safety will be assessed by cerebral magnetic resonance, neuropsychological examination and periprocedural transcranial Doppler measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients age > 18 years
* Patients with paroxysmal, or persistent/long-standing persistent AF according to the standard EHRA definition.
* Patients with symptomatic AF that is refractory to at least one antiarrhythmic medication.
* Absence of significant structural heart disease (dilated cardiomyopathy, hypertrophic cardiomyopathy, valvular heart disease, untreated coronary artery disease)

Exclusion Criteria:

* AF secondary to a reversible cause (i.e., thyreopathy, etc.) Indication for open-heart surgery (coronary artery bypass grafting, valve surgery, etc.)
* Severe left ventricle dysfunction that is clearly caused by some other cardiac disease (dilated cardiomyopathy, ischaemic heart disease, etc.) where the AF is clearly of secondary etiology
* Known severe pericardial and pleural adhesions (e.g., history of cardiac surgery)

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with symptomatic, drug-resistant, stand-alone, paroxysmal, persistent or long-standing persistent atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
efficacy - sinus rhythm | 1 year
  Number of patients with sinus rhythm, without detections of atrial arrhythmias (episodes longer than 30 seconds)

SECONDARY OUTCOMES:
periprocedural complications - surgery | 30 days after surgery
  conversion to sternotomy, bleeding, thromboembolic events, tamponade, haemothorax, pneumothorax, pleural effusion, pneumonia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tanaka K, Koga M, Lee KJ, Kim BJ, Park EL, Lee J, Mizoguchi T, Yoshimura S, Cha JK, Lee BC, Nakahara J, Suzuki N, Bae HJ, Toyoda K; CRCS-K Investigators and the SAMURAI Study Investigators. Atrial Fibrillation-Associated Ischemic Stroke Patients With Prior Anticoagulation Have Higher Risk for Recurrent Stroke. Stroke. 2020 Apr;51(4):1150-1157. doi: 10.1161/STROKEAHA.119.027275. Epub 2020 Feb 26. PMID 32098607